CLINICAL TRIAL: NCT06279234
Title: A Phase 1, Randomized, Double-Blind, Sponsor-Open, Placebo-Controlled Study to Assess the Safety, Tolerability, and Pharmacokinetics of Multiple Escalating Oral Doses of PF-06954522 in Adult Participants With Type 2 Diabetes Mellitus
Brief Title: A Study to Learn How Different Amounts of PF-06954522 Are Tolerated and Act in Adults With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: C4001002; NCT06279234 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2024-02-19; First posted 2024-02-28 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Obesity
Keywords: T2DM; Obesity; PF-06954522; Rosuvastatin; Midazolam; Omeprazole; DDI; C4001002
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Rosuvastatin Calcium; Midazolam; Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A (Experimental): Multiple doses of PF 06954522 or placebo daily for up to 8 weeks in adult participants with T2DM in up to 7 cohorts.
  Interventions: Drug: Placebo; Drug: PF-06954522
- Part B (Optional) (Experimental): Multiple doses of PF 06954522 or placebo daily for up to 8 weeks in non-diabetic adult participants with obesity in up to 3 cohorts.
  Interventions: Drug: Placebo; Drug: PF-06954522
- Part C (Optional) (Experimental): An 8-period multiple-dose assessment of the effect of PF-06954522 on rosuvastatin, midazolam, and omeprazole PK in healthy adult participants for up to 14 weeks in healthy adult participants.
  Interventions: Drug: Rosuvastatin; Drug: Midazolam; Drug: Omeprazole; Drug: PF-06954522

INTERVENTIONS:
Drug: Placebo — Oral tablet
  Arms: Part A; Part B (Optional)
Drug: Rosuvastatin — Oral tablet
  Arms: Part C (Optional)
Drug: Midazolam — Oral suspension
  Arms: Part C (Optional)
Drug: Omeprazole — Oral tablet
  Arms: Part C (Optional)
Drug: PF-06954522 — Oral tablet

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of multiple escalating oral doses of PF-06954522 in adult participants with inadequately controlled type 2 diabetes mellitus (T2DM) on metformin (Part A) and optionally in non-diabetic participants with obesity (Part B).

ELIGIBILITY:
Inclusion Criteria:

* Female participants of non-childbearing potential and males between the ages of 18 and 70 years, inclusive, at the time of signing the ICD.
* Part A only: Diagnosis of Diabetes - Participants enrolling with T2DM must have a clinical history of T2DM and be taking metformin monotherapy as their only anti-hyperglycemic treatment. Metformin dose must be at least 500 mg per day and must be stable, defined as no change in the treatment, including dose, for at least 2 months prior to the screening visit.

Part C only: Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.

* HbA1c

  * Part A only: For participants enrolling with T2DM: HbA1c ≥7.0% and ≤10.5% at screening (confirmed by a single repeat, if necessary).
  * Part B and C only: For participants enrolling as non-diabetic with obesity (Part B), or healthy (Part C): HbA1c <6.5% at screening.
* BMI

  * All participants must have a total body weight >50 kg (110 lbs).
  * Parts A and B only: Stable body weight, defined as <5 kg change (per participant report) for 90 days prior to screening
  * Part A only: For participants enrolling with T2DM: BMI ≥24.5 to ≤45.5 kg/m2.
  * Part B only: For participants enrolling as non-diabetic with obesity: BMI >30.5 to ≤45.5 kg/m2
  * Part C only: For participants enrolling as healthy: BMI 20-30.5 kg/m2
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICD and in this protocol.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, hepatic, psychiatric, neurological, dermatological, or allergic disease (including drug allergies but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).

  * Parts A and B only: Participants with T2DM (Part A) or obesity (Part B) are allowed. Participants who have chronic conditions other than T2DM and obesity (eg, hypercholesterolemia or hypertension) but are controlled by either diet or stable doses of 2 or fewer medications may be included (eg, a participant with hypercholesterolemia on appropriate treatment is eligible).
  * Any condition possibly affecting drug absorption (eg, prior bariatric surgery, gastrectomy, or any area of intestinal resection, active inflammatory bowel disease or pancreatic insufficiency).
  * History of HIV infection, hepatitis B, or hepatitis C; positive testing for HIV, HBsAg, or HCVAb. Hepatitis B vaccination is allowed.
* Diagnosis of type 1 diabetes mellitus or secondary forms of diabetes.
* Parts B and C only: Participants enrolling as non-diabetic with obesity (Part B) or healthy (Part C) may not have medical history of T2DM.
* Evidence or history of clinically significant cardiovascular disease. In particular, history of myocardial infarction, unstable angina, arterial revascularization, stroke, New York Heart Association Functional Class II IV heart failure, or transient ischemic attack within 6 months of screening.
* Any malignancy not considered cured (except basal cell carcinoma and squamous cell carcinoma of the skin); a participant is considered cured if there has been no evidence of cancer recurrence in the previous 5 years.
* Acute pancreatitis or history of chronic pancreatitis.
* Acute gallbladder disease.
* Parts A and B only: A response of 'yes' to question 4 or 5 or on any behavioral question on the C-SSRS at Screening or Day -1 in the study. In addition, participants deemed by the investigator to be at significant risk of suicidal or violent behavior should be excluded.
* Personal or family history of MTC or MEN2, or participants with suspected MTC per the investigator's judgement.
* Any medical or psychiatric condition including recent (within the past year) history of: suicidal ideation/behavior, major depressive disorder, schizophrenia, bipolar disorder; or laboratory abnormality or other conditions that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study
* Use of prescription or nonprescription drugs and dietary and herbal supplements that are BCRP, MDR1/P-gp, or OATP inhibitors is prohibited within 14 days or 5 half-lives (whichever is longer) prior to the first dose of study intervention; use of moderate or strong inhibitors or inducers of CYP3A, UGT1A1, or UGT1A3 is prohibited within 14 days plus 5 half-lives prior to the first dose of study intervention.

  * Part A and B: Use of certain concomitant medication that are unlikely to interfere with the study results may be allowed. However, use of prescription or nonprescription drugs and dietary and herbal supplements that are sensitive CYP1A2, CYP2C19, CYP3A, BCRP, MDR1/P-gp, OATP1B3, or UGT1A1 substrates is prohibited post Day -1.
  * Part C: Use of moderate or strong inhibitors or inducers of CYP2C19 are prohibited within 14 days plus 5 half-lives prior to the first dose of study intervention. Use of all other prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study intervention.
* Use of any prohibited prior/concomitant medication(s) or participant unwilling or unable to use a required concomitant medication(s).
* Previous administration of an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer).
* Known prior participation (ie, randomized and received at least 1 dose of study intervention) in a trial involving PF-06954522. Note that a given individual may only participate in a single cohort of this study.
* A positive urine drug screen at screening or admission. Participants who have been medically prescribed benzodiazepines and report the use of these drugs to the investigator at the screening visit may be allowed to participate if approved by the sponsor.
* Parts A and B only: Screening supine BP ≥160 mm Hg (systolic) or ≥100 mm Hg (diastolic) following at least 5 minutes of supine rest. If BP is ≥160 mm Hg (systolic) or ≥100 mm Hg (diastolic), the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility.

Part C only: Screening supine BP ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic) for participants <60 years; and ≥150/90 mm/Hg for participants ≥60 years old, following at least 5 minutes of supine rest. If systolic BP is ≥140 or 150 mm Hg (based on age) or diastolic ≥90 mm Hg, the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility.

- Screening 12-lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, baseline QTcF interval >450 ms, complete left bundle branch block, signs of an acute or indeterminate age myocardial infarction, ST-T interval changes suggestive of myocardial ischemia, second- or third- degree atrioventricular block, or serious bradyarrhythmias or tachyarrhythmias).

If QTcF exceeds 450 ms, or QRS exceeds 120 ms, the ECG should be repeated 2 more times and the average of the 3 QTcF or QRS values should be used to determine the participant's eligibility. Computer interpreted ECGs should be overread by a physician experienced in reading ECGs before excluding participants.

* Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study-specific laboratory and confirmed by a single repeat test if deemed necessary:

  * AST or ALT level ≥1.5 × ULN;
  * Total bilirubin level ≥1.5 × ULN; participants with an elevated total bilirubin consistent with Gilbert's Disease will have a direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is ≤ULN;
  * TSH > ULN;
  * Fasting C-peptide <0.8 ng/mL;
  * Serum calcitonin > ULN;
  * Amylase > ULN;
  * Lipase > ULN.
* Fasting blood glucose

  * Part A only: >270 mg/dL at screening or admission, confirmed by a single repeat test if deemed necessary.
  * Parts B and C only: >126 mg/dL at screening or admission, confirmed by a single repeat test if deemed necessary.
* Renal impairment as defined by an eGFR <75 mL/min/1.73m2. Confirmation of screening eGFR by a single repeat test is permitted, if deemed necessary.

  • Based upon participant age at screening, eGFR is calculated using the recommended CKD-EPI equations in Section 10.7.2 to determine eligibility (Screat-based formula).
* History of alcohol abuse or binge drinking and/or any illicit drug use or dependence within 6 months of Screening. Binge drinking is defined as a pattern of 5 (male) and 4 (female) or more alcoholic drinks in about 2 hours. As a general rule, alcohol intake should not exceed 14 units per week (1 unit = 8 ounces ([240 mL] beer, 1 ounce [30 mL] of 40% spirit or 3 ounces [90 mL] of wine).
* Prior use of a GLP-1R agonist within 6 months prior to screening or known intolerance to any GLP-1R agonist.
* Body weight exceeds the maximum capacity of the site's body weight scale, preventing accurate assessment of body weight.
* Part C only: History of hypersensitivity, intolerance, or allergic reaction associated with prior exposure to rosuvastatin, midazolam, or omeprazole.
* Part C only: Use of tobacco/nicotine containing products in excess of the equivalent of 5 cigarettes/day or 2 chews of tobacco/day.
* Investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-02-20 (Actual); Primary Completion 2025-04-11 (Actual); Study Completion 2025-04-11 (Actual)

PRIMARY OUTCOMES:
Number of Participants Reporting Adverse Events | Baseline through Week 14
Number of Participants with Clinically Significant Change From Baseline in Laboratory Abnormalities | Baseline through Week 14
Number of Participants With Clinically Significant Change From Baseline in Vital Signs | Baseline through Week 14
Number of Participants With Clinically Significant Change From Baseline in 12-Lead ECGs | Baseline through Week 14
Number of Participants with categorical scores on the Columbia Suicide Severity Rating Scale (C-SSRS) | Baseline through Week 14

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Part A: Days -1, 1, 14, 21 & 28. Days 2, 4, 7, 10, 17, 20, 24, 30. Part A & B: Days -1, 1, 28, 49 & 56. Days 7, 14, 21, 35, 42, 57 & 58. Part C: Period 3 Day 3 & Period 5 Day 28
Area Under the Curve from Time Zero to end of dosing interval (AUCtau) | Part A: Days -1, 1, 14, 21 & 28. Days 2, 4, 7, 10, 17, 20, 24, 30. Part A & B: Days -1, 1, 28, 49 & 56. Days 7, 14, 21, 35, 42, 57, 58. Part C: Period 3 Day 3 & Period 5 Day 28
Time to Reach Maximum Observed Plasma Concentration (Tmax) | Part A: Days -1, 1, 14, 21 & 28. Days 2, 4, 7, 10, 17, 20, 24 & 30. Part A & B: Day -1, 1 28, 49 & 56. Days 7, 14, 21, 35, 42, 57 & 58. Part C: Period 3 Day 3 & Period 5 Day 28
Plasma Decay Half-Life (t1/2) | Part A: Day -1, 1,14, 21 & 28. Days 2, 4, 7, 10, 17, 20, 24 & 30. Part A & B: Day -1, 1, 28, 49 & 56. Days 7, 14, 21, 35, 42, 57 & 58. Part C: Period 3 Day 3 & Period 5 Day 28
Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) | Part A: Day 28. Part A & B: Day 56
Percentage of Dose of PF-06751979 Excreted Unchanged in the Urine Over the Dosing Interval Tau (Aetau%) | Part A: Day 28. Part A & B: Day 56
Renal Clearance (CLr) | Part A: Day 28. Part A & B: Day 56

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Qps-Mra, Llc, South Miami, Florida

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4001002